CLINICAL TRIAL: NCT03131154
Title: A Phase 3, Randomized, Double-masked, Vehicle-controlled Trial to Evaluate the Safety and Efficacy of ADX-102 Ophthalmic Solution in Subjects With Non-infectious Anterior-uveitis.
Brief Title: SOLACE Trial - A Phase 3 Trial in Subjects With Non-infectious Anterior-uveitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-UV-005
Record Dates: First submitted 2017-04-04; First posted 2017-04-27 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2020-05

CONDITIONS: Non-infectious Anterior Uveitis
Keywords: reproxalap
MeSH Terms: interventions — reproxalap

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-102 Ophthalmic Solution (0.5%) (Experimental)
  Interventions: Drug: ADX-102 Ophthalmic Solution (0.5%)
- Vehicle of ADX-102 Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle of ADX-102 Ophthalmic Solution

INTERVENTIONS:
Drug: ADX-102 Ophthalmic Solution (0.5%) — ADX-102 Ophthalmic Solution (0.5%) administered for approximately four weeks.
  Other Names: Reproxalap
  Arms: ADX-102 Ophthalmic Solution (0.5%)
Drug: Vehicle of ADX-102 Ophthalmic Solution — Vehicle of ADX-102 Ophthalmic Solution administered for approximately four weeks.
  Other Names: Vehicle of Reproxlap
  Arms: Vehicle of ADX-102 Ophthalmic Solution

SUMMARY:
A Phase 3, randomized, double-masked, vehicle-controlled trial to evaluate the safety and efficacy of ADX-102 ophthalmic solution in Subjects with non-infectious anterior-uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥ 18 years and ≤ 85 years.
* Subjects with acute non-infectious anterior uveitis with onset of symptoms within the previous 2 weeks.
* Best corrected visual acuity (BCVA) better than or equal to 35 letters in the study eye and 65 letters in the non-study eye using ETDRS testing.

Exclusion Criteria:

* Have severe/serious ocular pathology in the study eye(s) which may preclude study completion, in the judgement of the Investigator.
* Active intermediate or posterior uveitis in the study eye(s).
* Previous anterior uveitis episode in the study eye ≤ 4 weeks prior to screening.
* Have participated in another investigational device or drug study within 30 days prior to screening.
* Participation in a prior ADX-102 study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - UAB Department of Ophthalmology, Birmingham, Alabama
  - Retinal Research Institute, Phoenix, Arizona
  - M&M Eye Institute, Prescott, Arizona
  - Walman Eye Center, Sun City, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - University of California, Irvine, Irvine, California
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Corneal Consultants of Colorado, Littleton, Colorado
  - Danbury Eye Physicians & Surgeons, Danbury, Connecticut
  - Levenson Eye Associates, Jacksonville, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - John Hopkins, Baltimore, Maryland
  - Valley Eye Physicians & Surgeons, Ayer, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Ocular Immunology & Uveitis Foundation, Waltham, Massachusetts
  - Oakland Ophthalmic Surgery, Birmingham, Michigan
  - Tauber Eye Center, Kansas City, Missouri
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - Bergstrom Eye Research, Fargo, North Dakota
  - Oregon Retina, LLP, Eugene, Oregon
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Retina and Uveitis Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ADX-102 Ophthalmic Solution (0.5%): ADX-102 administered for approximately 4 weeks
- Vehicle Ophthalmic Solution: Vehicle administered for approximately 4 weeks
Period: Overall Study
Arm/Group | ADX-102 Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
Started | 61 | 62
Completed | 37 | 33
Not Completed | 24 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADX-102 Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (15.8) | 47.8 (17.9) | 46.5 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 41 | 75
  Male | 27 | 21 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 22 | 49
  Not Hispanic or Latino | 34 | 40 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 48 | 98
  Black or African American | 8 | 10 | 18
  Asian | 0 | 1 | 1
  American Indian or Alaska Native | 1 | 0 | 1
  Unknown | 1 | 0 | 1
  Other | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 61 | 62 | 123
Height [Mean (Standard Deviation); unit: centimeters] | 167.09 (9.72) | 169.30 (9.57) | 168.2 (9.67)
Weight [Mean (Standard Deviation); unit: kilograms] | 85.95 (20.62) | 85.45 (21.98) | 85.70 (21.23)
Subjects with Bilateral Uveitis [Number; unit: participants]
  Right Eye | 25 | 23 | 48
  Left Eye | 30 | 34 | 64
  Both Eyes | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Meet Time to Clearance of Anterior Chamber Cells
Description: Time to clearance of anterior chamber cells was defined as the time from initiation of study drug to when a cell count of 0 was achieved and maintained (without cell count increases to >0) to Week 4 and without rescue or discontinuation due to rescue prior to Week 4. Anterior chamber cell count is the number of cells visible within the anterior chamber of the eye, measured using a slit lamp and following SUN (Standardization of Uveitis Nomenclature) where a cell count <1 is Grade 0 (absent) and a cell count of >50 is Grade 4+ (severe).
Time Frame: The efficacy assessment period was 4 weeks; baseline was defined as Day 1.
Population: Intent-to-treat population
Measure: Number; unit: Subjects
Arm/Group | ADX-102 Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 61 | 62
Subjects | 25 | 24
Statistical Analysis 1: Comparison: ADX-102 Ophthalmic Solution (0.5%) vs Vehicle Ophthalmic Solution; Test type: Other; Hazard Ratio (HR) = 1.129, 95% CI 2-sided [0.643 to 1.982] — Cox proportional hazards model

2. Post Hoc Outcome: Number of Subjects With Time to Clearance of Anterior Chamber Cells in Grade 1+ or Grade 2+ Subjects With a Baseline Anterior Chamber Cell Count > 10
Description: as for outcome 1
Time Frame: The efficacy assessment period was 4 weeks; baseline was defined as Day 1.
Population: Intent-to-treat population in grade 1+ or grade 2+ subjects with a baseline anterior chamber cell count > 10
Measure: Number; unit: Subjects
Arm/Group | ADX-102 Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 26 | 26
Subjects | 13 | 6
Statistical Analysis 1: Comparison: ADX-102 Ophthalmic Solution (0.5%) vs Vehicle Ophthalmic Solution; Test type: Other; Hazard Ratio (HR) = 2.619, 95% CI 2-sided [0.989 to 6.939] — Cox proportional hazards model

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately five weeks.
Arm/Group | ADX-102 Ophthalmic Solution (0.5%) | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/61 | 2/62
Other Adverse Events (participants affected / at risk) | 36/61 | 31/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADX-102 Ophthalmic Solution (0.5%) (N=61) | Vehicle Ophthalmic Solution (N=62)
Visual acuity reduced (Eye disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0 — The adverse event of suicide attempt was deemed by the Principal Investigator to be no related to drug.
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADX-102 Ophthalmic Solution (0.5%) (N=61) | Vehicle Ophthalmic Solution (N=62)
Uveitis (Eye disorders) | 7 | 7
Eye pain (Eye disorders) | 7 | 7
Visual acuity reduced (Eye disorders) | 3 | 6
Iridocyclitis (Eye disorders) | 4 | 3
Eye inflammation (Eye disorders) | 2 | 4
Vitreous floaters (Eye disorders) | 0 | 4
General Disorders and Administration Site Conditions (General disorders) | 13 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03131154/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03131154/SAP_002.pdf